CLINICAL TRIAL: NCT03949673
Title: Study to Evaluate Arthroplasty Specimens in the Phase 3 Fasinumab Program for Osteoarthritis of the Knee and Hip
Brief Title: Study to Evaluate Arthroplasty Specimens for Osteoarthritis of the Knee and Hip
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R475-OA-1816; 2018-001618-13 (EudraCT Number)
Record Dates: First submitted 2019-04-05; First posted 2019-05-14 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — fasinumab; Naproxen; Diclofenac; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Knee or Hip Joint Arthroplasty (Other): Patients with OA of the knee or hip who are participating in an ongoing fasinumab phase 3 parent study
  Interventions: Drug: Fasinumab; Drug: Naproxen; Drug: Diclofenac; Drug: Celecoxib; Drug: Placebo

INTERVENTIONS:
Drug: Fasinumab — Study drug will be administered in the parent study. Samples will be collected for participants who voluntarily elect to have knee or hip joint arthroplasty during the parent study
  Other Names: REGN475
Drug: Naproxen — Naproxen will be administered in the parent study. Samples will be collected for participants who voluntarily elect to have knee or hip joint arthroplasty during the parent study
Drug: Diclofenac — Diclofenac will be administered in the parent study. Samples will be collected for participants who voluntarily elect to have knee or hip joint arthroplasty during the parent study
  Other Names: ZORVOLEX
Drug: Celecoxib — Celecoxib will be administered in the parent study. Samples will be collected for participants who voluntarily elect to have knee or hip joint arthroplasty during the parent study
  Other Names: CELEBREX
Drug: Placebo — Matching Placebo will be administered in the parent study. Samples will be collected for participants who voluntarily elect to have knee or hip joint arthroplasty during the parent study

SUMMARY:
The objective of this exploratory study is to evaluate the cellular and connective tissue composition of joints from patients with Osteoarthritis (OA) who have been treated with fasinumab, compared with those treated with placebo or Non-steroidal anti-inflammatory drugs (NSAIDs).

ELIGIBILITY:
Key Inclusion Criteria:

* Previously randomized to R475-PN-1523 (NCT02683239), R475-OA-1611 (NCT03161093), or R475-OA-1688 (NCT03304379) and received at least 1 dose of study drug
* Notified the site that they are planning a knee or hip arthroplasty during the parent study between randomization and 24 weeks after the last dose of subcutaneous (SC) study drug
* Patient's surgeon/pathologist is willing to coordinate with the site regarding preparation, storage, and shipping of joint tissue samples collected during arthroplasty surgery

Exclusion Criteria:

* None

Note: Other protocol Inclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (15):
- United States (6):
  - Regeneron Research Site, Phoenix, Arizona
  - Regeneron Research Site, Littleton, Colorado
  - Regeneron Research Site, Jacksonville, Florida
  - Regeneron Research Site, Chicago, Illinois
  - Regeneron Research Site, Brooklyn, New York
  - Regeneron Research Site, New York, New York
- Regeneron Recruting SIte, Bialystok, Poland
- United Kingdom (8):
  - Regeneron Research Site, Reading, Berkshire
  - Regeneron Research Site, Glasgow, Lanarkshire
  - Regeneron Research Site, Romford, London City
  - Regeneron Research Site, Northwood, Middlesex
  - Regeneron Research Site, Hexham, Northumberland
  - Regeneron Research Site, Yaxley, Peterborough
  - Regeneron Research Site, Kenilworth, Warwickshire
  - Regeneron Research Site, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, EMA, PMDA, etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study only included participants that received at least 1 dose of study drug in one of the 3 parent studies: R475-PN-1523 (NCT02683239), R475-OA-1611 (NCT03161093), or R475-OA-1688 (NCT03304379).
Groups:
- Placebo: Placebo was administered in the parent studies; joint tissue samples for this study were collected for participants who voluntarily elected to have knee or hip joint arthroplasty during the parent studies
- Non-steroidal Anti-inflammatory Drug (NSAID): Non-steroidal anti-inflammatory drugs (NSAID) were administered in the parent studies; joint tissue samples for this study were collected for participants who voluntarily elected to have knee or hip joint arthroplasty during the parent studies
- Fasinumab: Fasinumab was administered in the parent studies; joint tissue samples for this study were collected for participants who voluntarily elected to have knee or hip joint arthroplasty during the parent studies
Period: Overall Study
Arm/Group | Placebo | Non-steroidal Anti-inflammatory Drug (NSAID) | Fasinumab
Started | 2 | 5 | 13
Completed | 2 | 5 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Arthroplasty analysis set: All subjects who are enrolled in this study, have histological evaluation data and is based on the treatment received in their parent study (as treated).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Non-steroidal Anti-inflammatory Drug (NSAID) | Fasinumab | Total
Number analyzed (Participants) | 2 | 5 | 13 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (7.8) | 60.2 (7.7) | 67.3 (8.2) | 64.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 7 | 12
  Male | 0 | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 5 | 12 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 2 | 5 | 12 | 19
    Other | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants by Degree of Synovial Lymphocytic Inflammation
Description: Inflammatory cells including lymphocytes, mast cells, neutrophils, and eosinophils were scored by presence and degree (None present, Slight/Mild, Moderate, Marked/Band).
Time Frame: Up to 24 weeks from the last dose of study drug in the parent study, an average of approximately 3 months
Population: Arthroplasty analysis set: All participants who are enrolled in this study, have histological evaluation data and is based on the treatment received in their parent study (as treated).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Non-steroidal Anti-inflammatory Drug (NSAID) | Fasinumab
Number analyzed (Participants) | 2 | 5 | 13
Participants
  None present | 0 | 2 | 3
  Slight/Mild | 0 | 2 | 5
  Moderate | 2 | 1 | 3
  Marked/Band | 0 | 0 | 2

2. Primary Outcome: Number of Participants by Degree of Cartilage Loss
Description: Microscopic articular features including degree of cartilage were evaluated and scored (Superficial Fibrillation, Deep fissuring, Loss to Tide Mark, Loss to Exposed Bone).
Time Frame: Up to 24 weeks from the last dose of study drug in the parent study, an average of approximately 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Non-steroidal Anti-inflammatory Drug (NSAID) | Fasinumab
Number analyzed (Participants) | 2 | 5 | 13
Participants
  Superficial Fibrillation | 0 | 1 | 2
  Deep fissuring | 1 | 0 | 0
  Loss to Tide Mark | 0 | 1 | 2
  Loss to Exposed Bone | 1 | 3 | 9

3. Primary Outcome: Number of Participants by Degree of Bony Changes
Description: Microscopic articular features including degree of bony changes were evaluated and scored (Normal, Sclerosis [Lamellar/Mixed], Subarticular Fracture/Collapse).
Time Frame: Up to 24 weeks from the last dose of study drug in the parent study, an average of approximately 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Non-steroidal Anti-inflammatory Drug (NSAID) | Fasinumab
Number analyzed (Participants) | 2 | 5 | 13
Participants
  Normal | 1 | 1 | 1
  Sclerosis (Lamellar/Mixed) | 1 | 2 | 7
  Subarticular Fracture/Collapse | 0 | 2 | 5

ADVERSE EVENTS:
Time Frame: Safety was not analyzed or collected specifically for this sub-study
Description: Participants followed screening and pre-randomization requirements of their parent study and if they decided to undergo a joint replacement during the parent study, they could consent to this substudy. Safety data were collected during the parent studies.
Arm/Group | Placebo | Non-steroidal Anti-inflammatory Drug (NSAID) | Fasinumab
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was anticipated to close in Feb 2021, but ended prematurely on 25 Aug 2020 (date of global last arthroplasty surgery for last subject enrolled) due to lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT03949673/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT03949673/SAP_001.pdf